CLINICAL TRIAL: NCT06028425
Title: A Phase 1 Study to Evaluate the Effect of Food on the Pharmacokinetics of LOXO-783 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Food on LOXO-783 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-PIK-22004; J4C-OX-JZUC (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LOXO-783 (Fasted State) (Experimental): LOXO-783 administered orally to participants who are in fasted state
  Interventions: Drug: LOXO-783
- LOXO-783 (Fed State - Low Fat Meal) (Experimental): LOXO-783 administered orally to participants who are on low fat meal
  Interventions: Drug: LOXO-783
- LOXO-783 (Fed State - High Fat Meal) (Experimental): LOXO-783 administered orally to participants who are on high fat meal
  Interventions: Drug: LOXO-783

INTERVENTIONS:
Drug: LOXO-783 — Administered orally.
  Other Names: LY3849524

SUMMARY:
The main purpose of this study is to measure how much of LOXO-783 is in the bloodstream and how the body handles and eliminates LOXO-783 when administered in fasting and fed states in healthy participants. The study will also evaluate the safety and tolerability of LOXO-783. Participation could last up to 63 days including screening period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status as defined by the absence of evidence of any clinically significant active or chronic disease
* Body mass index (BMI): 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive

Exclusion Criteria:

* Females who are lactating or of childbearing potential
* Clinically significant history of any drug sensitivity, drug allergy, or food allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LOXO-783 | Predose on Day 1 up to 96 hours postdose
  PK: Cmax of LOXO-783
PK: Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC [0-∞]) of LOXO-783 | Predose on Day 1 up to 96 hours postdose
  PK: AUC [0-∞] of LOXO-783

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Guo-Avrutin, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Fortrea Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No